CLINICAL TRIAL: NCT06076993
Title: Effectiveness of the BodyKind School-based Body Image Intervention: a Cluster Randomised Control Trial
Brief Title: Cluster Randomised Control Trial of the BodyKind Body Image Programme
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Dublin (Other)
Collaborators: Jigsaw, The National Centre for Youth Mental Health, Ireland (Unknown); Irish Research Council (Other); Be Real USA NFP (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UCDublin1
Record Dates: First submitted 2023-09-27; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-09

CONDITIONS: Body Image

STUDY DESIGN:
Intervention Model Description: This is a parallel two-arm cluster randomized controlled effectiveness trial. This pragmatic trial will be conducted in settings similar to the "real world" which will include use of a school setting, teacher-led delivery during classroom time, no strict exclusion criteria for students and comparison to routine lessons-as-usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BodyKind programme group (Experimental): The intervention group will receive the BodyKind body image programme. The four 50 minute lessons of the BodyKind programme will be delivered by teachers at a rate of 1 lesson per week over four consecutive weeks.
  Interventions: Behavioral: BodyKind programme
- Waitlist control (No Intervention): The waitlist control group will engage in classes as usual and will receive the BodyKind programme after data is collected.

INTERVENTIONS:
Behavioral: BodyKind programme — BodyKind is a four-session, teacher-led, school-based programme for adolescents aged 15-17 years. This programme was developed by a team of international experts in body image and incorporates empirically supported principles of cognitive dissonance (which involves publicly criticising body ideals) and self-compassion (which involves reappraising self-critical evaluations). BodyKind also contains a social activism component that aims to tackle appearance biases, discrimination and racism and promote greater inclusivity and compassion for others.
  Programme Outline Lesson 1. Appearance Bias Lesson 2. Self-compassion & social media Lesson 3. Compassion for others Lesson 4. Becoming agents of change Learning Objectives
  * To cultivate skills in awareness, mindfulness, non-judgement, reflection, conscientiousness, compassion
  * To decrease levels of body dissatisfaction and self-criticism
  * To improve levels of self-compassion, positive body image, psychological wellbeing
  Arms: BodyKind programme group

SUMMARY:
Body dissatisfaction, a primary risk factor for eating disorders, is prevalent among adolescents. Given increases in adolescent body dissatisfaction since the Covid-19 pandemic, there is a pressing need for universal body image interventions, particularly for older adolescents aged 15-17 years, as this is a peak time for the onset of adolescent body image concerns; however, currently there are no evidence-based body image programmes for this age group.

This cluster randomised control trial will evaluate the effectiveness of BodyKind, a four session, teacher led, mixed gender body image intervention for older adolescents that incorporates empirically supported principles of self-compassion, cognitive dissonance and social justice. The version of BodyKind culturally adapted for the Irish context will be evaluated in adolescents aged 15-17 years in fourth year in post-primary schools in Ireland. Primary outcomes of body dissatisfaction, body appreciation and psychological wellbeing, in addition to secondary outcomes of body ideal internalisation, self-compassion and compassion for others will be assessed at pre, post and 2 month follow up in intervention groups (who receive the BodyKind programme) and waitlist controls.

DETAILED DESCRIPTION:
Design:

This pragmatic trial will be conducted in settings similar to the "real world" which will include use of a school setting, teacher-led delivery during classroom time, no strict exclusion criteria for students and comparison to routine lessons-as-usual. Data collection time points will be selected to align with school academic calendars and will be conducted at pre, post and two month follow up. Schools will be randomly allocated to an intervention group (who receive the BodyKind programme) or a waitlist control. Participants in intervention and waitlist groups complete measures at the same timepoints, and those in the waitlist control will receive BodyKind after all assessments are completed. A mixed methods evaluation of implementation quality will also be conducted to understand 'why' programme outcomes were observed and inform efforts to optimise programme delivery in schools in the future.

Randomization:

Prior to randomization, schools will be stratified based on school categorization (e.g., co-educational/ single sex girls/ single sex boys), size (i.e., estimated number of students in Transition Year available to participate) and location (i.e., urban/rural categorisation) to ensure the gender and geographical location of participants in each treatment group will be closely balanced. Shortlisted schools will be then randomly allocated to condition by the primary researcher using a computer-generated minimisation procedure. Minimisation is a method of randomisation that allocates participants to the treatment group that best maintains balance in prognostic factors (e.g., gender balance across condition). The first participant is allocated a treatment at random. Each subsequent participants' allocation is determined by what treatment allocation would lead to better balance between the groups in the variables of interest. Minimisation ensures excellent balance across treatment groups and is desirable when there are strong prognostic factors (e.g., gender) and modest treatment effects. Shortlisted* stratified schools will be allocated using covariate-constrained randomisation, a type of minimisation randomisation, for a two arm cluster randomized control trial, with the R statistical package cvcrand (https://cran.r-project.org/web/packages/cvcrand/cvcrand.pdf). Allocation of schools to experimental/waitlist treatment groups will be constrained by a.) the number of boys in TY in each school, b.) the number of girls in TY, and c.) the school's location categorisation (urban/rural). Schools that drop out will be replaced by schools on the waitlist based on minimisation or replacement by same category to same allocation (e.g., if an urban school drops out/fails to sign principal consent form they will be replaced by an urban school on the waitlist and to the allocation assigned to that urban school).

Data collection procedures:

Recruitment will occur at the school level. Schools will be recruited via emails (Educator School Centre's Ireland's mailing list and cold call invitations), teacher training events and advertisement on social media & website pages. Schools will be selected on the basis of (1) their expressed interest and (2) their fit with recruitment criteria.

Shortlisted schools registering interest and meeting these criteria that decline to participate after initial contact will be replaced by the next school from the waitlist of eligible schools who registered interest with the researcher. Schools will receive a €200 financial honorarium for participating.

Sample size:

The aim is to recruit 600 students aged 15-17 years in 4th year who attend second-level schools in Ireland. The aim is also to recruit 1-2 second-level teachers per school, from 12-28 schools, to deliver the BodyKind programme to adolescents.

Sample size rationale An RMASS power analysis (http://www.rmass.org/RMASS_Manual.pdf) based on parameters; small Cohen's d effect size of .2, power .80, alpha .05, indicates that 504 students are required. To account for natural attrition and unanticipated events that reduce participant numbers (e.g., student absence due to illness) in RCTs, approximately 20% (n=100) more participants will be recruited giving a total N=600. A systematic review of consent procedures and participation rates reported that the average consent rate for active parental consent was 65.5% (range: 11-100%). The average number of students in TY in schools in Ireland is 140; therefore, allowing for a 65% response rate would indicate that a minimum of 8 schools would be required to obtain a sample size of 600. However, a recent pilot trial of a self-compassion body image intervention in Ireland recruited an average of 25 TY students per school using opt in parental consent (4 schools, N=100), indicating that n=24 schools would be required to attain a sample size of 600. Given the variability in class size in Transition Year and range in consent rates for active parental consent the investigators will seek to recruit within this range until sample size of 600 is met. To guard against drop out at a cluster level the investigators will aim to oversample and recruit at least 12 schools and a maximum of 28 schools.

Hypotheses:

The hypotheses are

1. Compared to participants in the waitlist control, participants who receive the BodyKind programme will experience statistically significant increases in a.) body appreciation, psychological wellbeing, self-compassion and compassion for others and b.) significant decreases in body dissatisfaction and body ideal internalisation from pre- to post-intervention.
2. Changes will be maintained in experimental groups at a 2-month follow up.
3. Changes in body appreciation and body dissatisfaction will be mediated by self-compassion, compassion for others and body ideal internalisation. No a-priori assumptions about the directionality of effects will be made.
4. Changes in body appreciation, body dissatisfaction and psychological wellbeing will be moderated by appearance related social media use, appearance teasing, gender, baseline body appreciation, body dissatisfaction, psychological wellbeing and implementation quality. There are no a-priori assumptions about the directionality of effects.
5. The programme will be considered acceptable and feasible by adolescents and teachers
6. The programme can be implemented with high fidelity by teachers

Data analysis plan:

Prior to conducting inferential statistics, data will be screened for missingness, outliers, normality and model assumptions. Data will be summarised graphically and by using descriptive statistics.

H1. Generalised linear mixed effects models (GLMM) will be used to determine change on outcome measures. Primary analysis will compare measures at time one (baseline) and two (post-intervention), to identify fixed effects of the intervention. Potential clustering effects will be examined and accounted for at the school level. The model will include 2 main effects (1. Repeated measures effect of time and 2. Between subjects effect of condition) and one two way interaction (time*condition). Gender effects will also be considered. With gender in the model will have three main effects and corresponding two-way and three-way interactions.

H2. Secondary analyses will examine data from time 3 (follow-up) to see if the intervention condition has maintained hypothesised changes in dependent variables. Investigators will also assess the proportion of within-group and between-group variance by calculating the ICC. As complex models can fail to converge, if investigators encounter convergence issues in our models, investigators may consider dropping the random effect accounting for the smallest proportion of between-group variance. *Note: If the recruitment target (n=600) is not met, a different statistical analytic technique, 2 (condition; experimental, control) x 3 (time; pre, post, follow up) mixed factorial ANOVA will be used. This can detect small effects, but not clustering effects, in a sample size of 238 participants, according to a MorePower analysis. Post-hoc planned comparisons will be conducted using t-tests to examine changes within groups (intervention vs control) at different time points.

H3. Mediation analyses will investigate whether changes in body ideal internalisation, self-compassion and compassion for others mediate change in body dissatisfaction and positive body image from T1 to T2.

H4. Moderation analyses will investigate whether appearance related social media use, appearance teasing, gender, school type, baseline body appreciation, body dissatisfaction, psychological wellbeing and implementation quality moderate changes from T1 to T2.

H5. Descriptive statistics will be used to assess teacher fidelity ratings

ELIGIBILITY:
Inclusion Criteria:

* Schools will be eligible if

  1. they are a second-level school in Ireland that offers the Transition Year (TY) programme to students
  2. will deliver the intervention as part of their curriculum to students in TY
  3. teaching staff are willing to complete the 2.5-hour BodyKind teacher training programme.

Students will be eligible if

* they are in TY in a second-level school in Ireland and are aged 15-17 years
* If their parent consents to their participation AND if they provide a signed assent form .

Teachers will be eligible if

* They are qualified secondary school teacher
* They agree to complete the BodyKind teacher training
* Return a signed informed consent form

Exclusion Criteria:

* Schools will be excluded if

  * they are not a second-level school in Ireland or if they do not offer the TY programme to students
  * will not deliver the intervention as part of their curriculum to students in TY
  * teaching staff are not willing to complete the 2.5-hour BodyKind teacher training programme.

Students will be excluded if

* they are not in TY in a second-level school and are not aged 15-17 years
* If parental consent has not been obtained OR if they fail to sign a participant assent .

Teachers will be excluded if

* They are not qualified secondary school teacher
* They do not agree to complete the BodyKind teacher training
* Do not return a signed informed consent form

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Body Appreciation | 1 week pre-intervention, 1 week post-intervention, 2 month post intervention follow up
  Body Appreciation Scale-2 is a 10-item scale. Responses to items such "I feel good in my body" are indicated on a 5-point Likert Scale (1-5), with higher scores indicating higher levels of body appreciation (Min-Max: 10-50). BAS-2 demonstrates good validity and reliability among international adolescent samples
Body Dissatisfaction | 1 week pre-intervention, 1 week post-intervention, 2 month post intervention follow up
  Body Satisfaction Visual Analogue Scales Items from the appearance/weight subscales of the Eating Disorder Examination Questionnaire will be adapted as 10-point visual analogue scales (VAS) to assess state body satisfaction with various aspects of appearance. Participants will use a 10-point slider 0 (not at all satisfied) and 10 (very satisfied) to rate how satisfied they feel with their body shape, weight, and size. Participants will also rate their satisfaction with height, muscle mass/tone and overall appearance. A mean score from the six appearance dimensions will be calculated, with higher scores representing higher state body satisfaction. This approach has been shown to have good convergent validity with the Eating Disorder Inventory Body Dissatisfaction Subscale in adolescents (r = .62). Higher scores indicate higher body satisfaction. (Min-Max score: 6-60]
Psychological wellbeing | 1 week pre-intervention, 1 week post-intervention, 2 month post intervention follow up
  The Five-Item World Health Organisation Wellbeing Index is a unidimensional scale that measures emotional wellbeing using five positively worded items. Participants indicate the extent to which positive feelings, such as "I have felt calm and relaxed" were experienced over the last two weeks, using 6-point Likert scales ranging from 0 (not present) to 5 (constantly present). Raw scores are transformed to a score from 0 (worst thinkable well-being) to 100 (best thinkable well-being) with scores <50 suggesting poor emotional well-being.The WHO-5 has been validated for use with adolescents and has adequate validity as an outcome measure in clinical trials

SECONDARY OUTCOMES:
Self-compassion | 1 week pre-intervention, 1 week post-intervention, 2 month post intervention follow up
  The Self-Compassion Scale for Youth is a shortened and modified version of the Self-Compassion Scale developed for use with adolescent populations. The SCS-Y is a 14-item scale that contains subscales for the aspects of compassion; self-kindness, self-judgement, common humanity, isolation, mindfulness and over identification. Participants respond to items such as "When I feel frustrated or disappointed, I think about it over and over again." on 5-point Likert scales ranging from 1 (never) to 5 (always). Negatively worded items are reverse coded. Higher scores indicate higher levels of self-compassion [Min-Max scores: 14-70]. The SCS-Y has been validated among adolescents aged 12-17 years, where mean scores range between 1.0-2.49 (low), 2.5-3.5 (moderate), and 3.51-5.0 (high) and demonstrated good levels of internal consistency with Cronbach's alpha of >=.82 for each subscale.
Body ideal internalization | 1 week pre-intervention, 1 week post-intervention, 2 month post intervention follow up
  Internalization-General subscale of the Sociocultural Attitudes Towards Appearance Scale-3 will be used to assess internalization of social media ideals. Items were adapted to social media by substituting the words "social media" into item stems e.g. "I would like my body to look like people on social media". The five-item scale is measured using five-point Likert scales ranging from 1 (definitely disagree) and 5 (definitely agree). Negatively worded items are reversed coded and items are averaged to yield a mean score, with higher scores indicating greater body ideal internalization (Min-Max Score: 5-25). The original scale has been shown to be a reliable in adolescent girls and boys and the adapted scale has been found demonstrate good psychometric properties and good levels of internal consistency, ranging from α = 0.75 among male, and α = 0.84 among female adolescents
Appearance related social media use | 1 week pre-intervention, 1 week post-intervention, 2 month post intervention follow up
  The Appearance-Related Social Media Consciousness Scale is a 13-item scale that captures the extent to which individuals' thoughts and behaviours reflect ongoing awareness of whether they might look attractive to a social media audience. Given that appearance-related use is a more important predictor of body dissatisfaction compared with general/non-visual social media use, this measure is important to include. Items such as "I think about how specific parts of my body will look when people see my pictures on social media" are measured using 7-point Likert scales ranging from 1 (Never) to 7 (Always). Higher scores indicate higher levels of consciousness about appearance-related social media use (Min-Max score: 13-91) ASMC scores demonstrate strong internal consistency, convergent and incremental validity, and test-retest reliability in adolescent boys and girls
Compassion towards others | 1 week pre-intervention, 1 week post-intervention, 2 month post intervention follow up
  The Compassion Towards Others Action Subscale of the Compassionate Engagement and Action Scales Youth, measures compassion in adolescents. The 4-item action orientation competency subscale focuses specifically on actions aimed to prevent and alleviate distress/suffering in others, such as "When others are distressed or upset by things, I am kind and supportive to them". Participants respond using 10-point Likert scale from 0 (never) to 10 (always) with higher scores indicating higher compassionate action orientations towards others (Min-Max score: 0-40). This subscale shows good internal consistency with alpha values across items ranging between α=.84-.88 in adolescent boys and girls.

OTHER OUTCOMES:
Teacher fidelity | 1 week post intervention
  Teachers will complete a checklist at the end of each lesson indicating the extent to which they covered key aspects of the lessons. Teachers are required to cover 7 key learning objectives for each of the four lessons. Teachers indicate the number of key learning objectives they covered in each class delivered (1= Yes, 0=No). Higher scores indicate that more key learning objectives were covered by the teacher, thereby indicating higher levels of fidelity to the programme. (Min-Max score: 0-28)

CONTACTS AND LOCATIONS:
Overall Officials: Ciara Mahon, PhD, Principal Investigator — University College Dublin
Locations (1):
- University College Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
According to Article 9 of the GDPR, this research will involve the collection of special category data as it relates to a "person's ethnicity or racial origin, political opinions or religious or philosophical beliefs, health, genetic data, biometric data, sexual life and/or orientation, trade union membership". Given the sensitive and possibly identifying nature of the data, data cannot be publicly archived. In accordance with UCD's data retention policy, all data gathered for research will be stored in electronic form for five years from the end of the project, after which, data will be deleted.
  Although raw data cannot be publicly archived, all manuscripts will be submitted to open access journals. All studies will also be pre-registered on open platforms such as OSF (https://osf.io/) and on the discipline specific, Psychology Preprint Service 'PsyArXiv' (https://psyarxiv.com/) to ensure openness and transparency.

REFERENCES:
- [Background] Roy A, Bhaumik DK, Aryal S, Gibbons RD. Sample size determination for hierarchical longitudinal designs with differential attrition rates. Biometrics. 2007 Sep;63(3):699-707. doi: 10.1111/j.1541-0420.2007.00769.x. PMID 17825003
- [Background] Blom-Hoffman J, Leff SS, Franko DL, Weinstein E, Beakley K, Power TJ. Consent Procedures and Participation Rates in School-Based Intervention and Prevention Research: Using a Multi-Component, Partnership-Based Approach to Recruit Participants. School Ment Health. 2009 Mar 1;1(1):3-15. doi: 10.1007/s12310-008-9000-7. PMID 19834586
- [Background] Tylka TL, Wood-Barcalow NL. The Body Appreciation Scale-2: item refinement and psychometric evaluation. Body Image. 2015 Jan;12:53-67. doi: 10.1016/j.bodyim.2014.09.006. Epub 2014 Oct 21. PMID 25462882
- [Background] Durkin SJ, Paxton SJ. Predictors of vulnerability to reduced body image satisfaction and psychological wellbeing in response to exposure to idealized female media images in adolescent girls. J Psychosom Res. 2002 Nov;53(5):995-1005. doi: 10.1016/s0022-3999(02)00489-0. PMID 12445589
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Neff KD, Bluth K, Toth-Kiraly I, Davidson O, Knox MC, Williamson Z, Costigan A. Development and Validation of the Self-Compassion Scale for Youth. J Pers Assess. 2021 Jan-Feb;103(1):92-105. doi: 10.1080/00223891.2020.1729774. Epub 2020 Mar 3. PMID 32125190
- [Background] Thompson JK, van den Berg P, Roehrig M, Guarda AS, Heinberg LJ. The sociocultural attitudes towards appearance scale-3 (SATAQ-3): development and validation. Int J Eat Disord. 2004 Apr;35(3):293-304. doi: 10.1002/eat.10257. PMID 15048945
- [Background] Gordon CS, Rodgers RF, Slater AE, McLean SA, Jarman HK, Paxton SJ. A cluster randomized controlled trial of the SoMe social media literacy body image and wellbeing program for adolescent boys and girls: Study protocol. Body Image. 2020 Jun;33:27-37. doi: 10.1016/j.bodyim.2020.02.003. Epub 2020 Feb 18. PMID 32086189
- [Background] Choukas-Bradley S, Nesi J, Widman L, Galla BM. The Appearance-Related Social Media Consciousness Scale: Development and validation with adolescents. Body Image. 2020 Jun;33:164-174. doi: 10.1016/j.bodyim.2020.02.017. Epub 2020 Mar 17. PMID 32193170
- [Background] Henje E, Rindestig FC, Gilbert P, Dennhag I. Psychometric validity of the Compassionate Engagement and Action Scale for Adolescents: a Swedish version. Scand J Child Adolesc Psychiatr Psychol. 2020 Jul 18;8:70-80. doi: 10.21307/sjcapp-2020-007. eCollection 2020. PMID 33520779
- [Background] Walton H, Spector A, Tombor I, Michie S. Measures of fidelity of delivery of, and engagement with, complex, face-to-face health behaviour change interventions: A systematic review of measure quality. Br J Health Psychol. 2017 Nov;22(4):872-903. doi: 10.1111/bjhp.12260. Epub 2017 Aug 1. PMID 28762607
- [Background] Gattario KH, Frisen A. From negative to positive body image: Men's and women's journeys from early adolescence to emerging adulthood. Body Image. 2019 Mar;28:53-65. doi: 10.1016/j.bodyim.2018.12.002. Epub 2018 Dec 21. PMID 30583277
- [Background] Kurz M, Rosendahl J, Rodeck J, Muehleck J, Berger U. School-Based Interventions Improve Body Image and Media Literacy in Youth: A Systematic Review and Meta-Analysis. J Prev (2022). 2022 Feb;43(1):5-23. doi: 10.1007/s10935-021-00660-1. Epub 2021 Dec 28. PMID 34962632
- [Derived] Mahon C, Hamburger D, Webb JB, Yager Z, Howard E, Booth A, Fitzgerald A. Protocol of a cluster randomised trial of BodyKind: a school-based body image programme for adolescents. BMC Public Health. 2023 Nov 14;23(1):2246. doi: 10.1186/s12889-023-17002-x. PMID 37964252